CLINICAL TRIAL: NCT06164210
Title: Investigation of the Effect of Snoezelen-Based Occupational Therapy Intervention on Sleep and Behavioral Problems in 18-36 Months Children at Risk of Autism
Brief Title: Effect of Snoezelen-Based Occupational Therapy Intervention on Sleep and Behavior Problems in Infant at Risk of Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yusuf Islam Degerli, Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-177
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder; Sleep Disorder; Behavior Problem
Keywords: autism; behavioral problem; sleep disorder; sensory integration; Multi-sensory room
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Wake Disorders; Mental Disorders; Autistic Disorder; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Sensory Integration Intervention Group (Experimental): Conventional Sensory Integration Intervention Based on Sensory Processing Theory, sensory integration intervention increases a childs ability to process and integrate sensory information and thus create more organized and adaptive behaviors. Sensory-enriched environments use fun interactive games and activities. Sensory integration intervention is carried out by creating an intervention program to create, understand, and eliminate the deficiency of the sensory process.
  A conventional sensory integration intervention two sessions (per sessions 45 minutes) a week, was planned for 18-35-month-old infants at risk of ASD in both groups participating in the study. Session planning and activity selection were based on TSP-2 results. In particular, the occupational therapist supported the infant's active participation in the activities.
  Interventions: Behavioral: Snoezelen-Based Occupational Therapy Intervention Group
- Snoezelen-Based Occupational Therapy Group (Active Comparator): Snoezelen- Based Occupational Therapy Intervention Different from sensory integration interventions, Snoezelen interventions are environments with all sensory stimuli, such as auditory, visual, tactile, gustatory, olfactory, and vestibular stimuli, in the same environment and where therapeutic guidance and commands are not given to the individual. These interventions aim to reduce agitation, depression, and aggression in individuals and increase daily living activities, functional performance, and well-being. Psychiatric clinics, schools, rehabilitation centers, and occupational therapy clinics are some places where it is used. Some materials found in Snoezelen rooms are bubble tubes, fiber optic light cables, projectors, vibrating massagers, light tactile stimulation materials, aromatic scent emitting devices, music sets, and relaxing music and swings.
  Interventions: Behavioral: Snoezelen-Based Occupational Therapy Intervention Group

INTERVENTIONS:
Behavioral: Snoezelen-Based Occupational Therapy Intervention Group — Snoezelen- Based Occupational Therapy Intervention Different from sensory integration interventions, Snoezelen-based interventions are environments with all sensory stimuli, such as auditory, visual, tactile, gustatory, olfactory, and vestibular stimuli, in the same environment and where therapeutic guidance and commands are not given to the individual. These interventions aim to reduce agitation, depression, and aggression in individuals and increase daily living activities, functional performance, and well-being. Psychiatric clinics, schools, rehabilitation centers, and occupational therapy clinics are some places where it is used. Some materials found in Snoezelen rooms are bubble tubes, fiber optic light cables, projectors, vibrating massagers, light tactile stimulation materials, aromatic scent emitting devices, music sets, and relaxing music and swings.
  Other Names: Snoezelen; multi-sensory

SUMMARY:
Objective: Sleep and behavioral problems are common in infants at risk of autism. This study aims to examine the effect of Snoezelen-Based Occupational Therapy intervention on sleep and behavioral problems in infants at risk of autism. Design: Twenty-four infants (15 boys, 9 girls) at risk for autism were randomized to the intervention group (n = 12; 28.33 ± 6.52 months) and the control group (n = 9; 30.11 ± 5.20 years). The intervention group received Snoezelen-Based Occupational Therapy intervention in addition to the conventional 8-week sensory integration intervention, while the control group received only the conventional sensory integration intervention. Both groups assessed sleep and behavioral problems using the Brief Infant Sleep Questionnaire (BİSQ) and the Vineland Social-Emotional Early Childhood Scale (VSEES) pre and post eight weeks of intervention.

DETAILED DESCRIPTION:
Introduction Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by social interaction, social communication, and repetitive behavioral problems associated with sensory processing problems (SPP) that occur before the age of 3, according to The Diagnostic and Statistical Manual of Mental Disorders classification system (DSM-5). Early symptoms of ASD are characterized by limited social participation, inadequate performance in gestures, inability to initiate or maintain interactions with others, and repetitive movements. These symptoms are used as criteria for the diagnosis of ASD. However, in addition to the symptoms used as criteria, parents reported that they observed behavioral problems such as tantrums, senseless fear, and sleep problems in their children at risk for ASD more than in children with typical development. These additional symptoms observed by parents are also used as diagnostic criteria. Moreover, after eating problems, sleep problems, and SPP, tantrums and challenging behaviors are the most difficult for parents.

Sleep problems are 40% to 80% more common in ASD than in typically developing children. In children with typical development, this rate is between 25% and 40%. Sleep problems seen in ASD can be categorized under various headings. These include delayed falling asleep, sleep refusal, decreased sleep time, frequent awakenings, and bedtime resistance. The reason for the high prevalence of sleep problems in ASD is still unclear. Biological, genetic, intrinsic-motivational, behavioral, and sensory problems are thought to play a role.

The studies show that behavioral symptoms can cause sleep problems and that insufficient sleep triggers core behavioral ASD symptoms such as tantrums, aggression, and social communication difficulties. It is reported that sleep and behavioral problems are mutually triggering factors in ASD. In more detail, SPP may also cause sleep and behavior problems due to intrinsic-behavioral problems.

SPP is observed in more than 90% of children with ASD. According to DSM-5, SPP includes hyper- or hypo-reactive responses to sensory stimuli. Inappropriate responses to stimuli from the environment and the body cause behavioral problems. Sensory sensitivity causes problems in maintaining and sustaining calm and appropriate behavior toward the environment. Studies focusing on the relationship between ASD and sleep suggest that children with ASD who have problems with sensory reactivity, sensory seeking, and filtering incoming stimuli may have sleep disorders. In other words, behavioral problems caused by certain sensory stimuli can be seen as self-harm, aggression, and sleep problems. Sensory integration interventions in SPP aim to provide the infant with controlled and meaningful sensory experiences and accurate environmental responses. Sensory processing interventions are based on models such as sensory integration and snoezelen-based programs that incorporate neuroplasticity and engagement. Studies suggest deep pressure, vestibular, and tactile stimuli will help release endorphins and serotonin and increase perceived sleep quality and calmness in sensory-based sleep disorders.

Snoezelen-based interventions, in which sensory stimuli are experienced in intense and multiple ways, are generally used to reduce stress and depression and provide a sense of relaxation. Snoezelen-based interventions are used to relax individuals in various diagnostic groups, such as dementia and mental retardation, and to reduce agitation, depression, and aggression levels. In studies on ASD children, snoezelen-based interventions have improved social skills and decreased self-harm behaviors. It is stated that it positively affects sleep quality regarding its impact on sleep problems, but the evidence is insufficient.

In light of the literature, this study aimed to examine the effect of Snoezelen-Based Occupational Therapy intervention on sleep and social-emotional behavior problems in infant with ASD risk.

Materials and Methods This study was planned as a randomized controlled trial to examine the effect of Snoezelen-Based Occupational Therapy intervention on sleep and behavioral problems of infants at risk of ASD. The study was approved by the Health Sciences University Non-Interventional Research Ethics Committee with file number 2022-177. Before the study, the parents of the children were informed about the study and written informed consent was obtained from the parents. The study was carried out in a state occupational therapy clinic.

Participants Inclusion criteria were (1) volunteering to participate in the study, (2) having a chronological age between 18-35 months, (3) checking yes in at least three of the 23 questions in the modified Modified Early Childhood Autism Screening Scale (M-CHAT), and (4) having a definite difference in at least one sensory domain according to the results of the early childhood sensory questionnaire. Exclusion criteria were (1) having any chronic disease that could affect the study (orthopedic, epileptic, etc.) and (2) receiving or having received intervention than sensory integration intervention (Speech and Language Therapy, Special Education, etc.). 24 participants were randomly assigned to the intervention (n=12) and control group (n=12) using a computer-generated randomization technique. During the intervention, 3 infants dropped out of the study (change of location=1 and starting additional intervention=2). The study was completed with 12 infants in the intervention group and 9 infants in the control group.

Design

Data Collection Tools The Brief Infant Sleep Questionnaire (BISQ); and the Vineland Social-Emotional Early Childhood Questionnaire (VSEES); were administered by the second author to assess pre-intervention sleep patterns and adaptive behaviors in daily life. The Early Childhood Sensory Profile of Infancy 2 Questionnaire was also used to determine the content of the intervention in the snoezelen-based room.

Modified Early Childhood Autism Screening Scale (M-CHAT)

The M-CHAT, a screening tool suitable for detecting infant ASD symptoms, was developed by Robins et al.. In the test consisting of twenty-three questions, all questions are answered by the parents. In the validity study, the reliability of 23 questions of the M-CHAT was found to be high (α = 0.85). Internal reliability was found to be adequate for the 23 items and six critical items (α = 0.87 and α = 0.85, respectively). The sensitivity and selectivity of the test were 0.99 and 0.94, respectively.

Toddler Sensory Profile 2 (TSP-2)

The TSP-2 is a standardized scale that assesses sensory processing ability and its impact on activities of daily living using caregiver observations of children aged 7-36 months. Questions in the TSP-2 are divided into five sensory processing sections (Auditory, Visual, Vestibular, Tactile, and Oral Sensory Processing) or four quadrants (Low Recording, Sensory Searching, Sensory Sensitivity, and Sensory Avoidance). Caregivers reports behavior frequency in each item question on a 5-point Likert scale ranging from 1 (almost always) to 5 (almost never). Turkish validity and reliability were conducted. The TSP-2 shows high test-retest reliability (ICC = 0.95) and very good internal consistency for all domains.

Brief Infant Sleep Questionnaire (BISQ)

The scale developed assesses whether the infant/child has a sleep problem and the level of sleep with seven parameters. These seven parameters are: 1. Sleep onset time, 2. Time to fall asleep, 3. Frequency of nighttime awakenings, 4. Nighttime insomnia duration, 5. Nighttime sleep duration, 6. Daytime sleep duration, 7. Total sleep duration. Turkish adaptation, validity, and reliability study were conducted in 2011, and a positive, moderate to strong (0.35-0.85) and significant (0.001) correlation was found between the pre-test and post-test.

Vineland Social-Emotional Early Childhood Scale (VSEES) Sparrow developed VSEES to assess childrens social-emotional development from birth to 5 years and 11 months. The internal consistency coefficients of the scale, which was adapted into Turkish and the validity and reliability study conducted, were determined as 0.60 in the verbal relationship dimension of the interpersonal relations subscale, 0.52 in the social communication subscale, 0.63 in the play and leisure time subscale, and 0.82 in the coping and adaptation subscale. In the total scale, the internal consistency coefficient was 0.87.

Intervention

Conventional Sensory Integration Intervention Based on Sensory Processing Theory, sensory integration intervention increases a child's ability to process and integrate sensory information and thus create more organized and adaptive behaviors. Sensory-enriched environments use fun interactive games and activities. Sensory integration intervention is carried out by creating an intervention program to create, understand, and eliminate the deficiency of the sensory process.

A conventional sensory integration intervention two sessions (per sessions 45 minutes) a week, was planned for 18-35-month-old infants at risk of ASD in both groups participating in the study. Session planning and activity selection were based on TSP-2 results. In particular, the occupational therapist supported the infants active participation in the activities. The necessary sensory stimuli (proprioceptive, vestibular, tactile, etc.) were presented through interactive play.

Snoezelen-Based Occupational Therapy Intervention

In the intervention group, infants received Snoezelen-Based Occupational Therapy intervention twice a week, each session lasting 30 minutes, in addition to 8 weeks of traditional sensory integration intervention. This intervention was planned according to the sensory profiles of the infants. The swing, music system, aromatic scents and tactile tools in the room were added according to the differences in the sensory profiles of the infants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were (1) volunteering to participate in the study, (2) having a chronological age between 18-35 months, (3) checking yes in at least three of the 23 questions in the modified Modified Early Childhood Autism Screening Scale (M-CHAT), and (4) having a definite difference in at least one sensory domain according to the results of the early childhood sensory questionnaire.

Exclusion Criteria:

* Exclusion criteria were (1) having any chronic disease that could affect the study (orthopedic, epileptic, etc.) and (2) receiving or having received intervention than sensory integration intervention (Speech and Language Therapy, Special Education, etc.).

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Investigation of the change in sleep quality with Brief Infant Sleep questionnaire (BİSQ) in the intervention group receiving Snoezelen-Based Occupational Therapy training in 8 weeks | Baseline and Week 8
  Brief Infant Sleep questionnaire (BİSQ):
  The scale assesses whether the infant/child has sleep problems and the level of sleep with seven parameters. These seven parameters are: 1. sleep onset time, 2. time to fall asleep, 3. frequency of nighttime awakenings, 4. duration of insomnia at night, 5. duration of nighttime sleep, 6. duration of daytime sleep, 7. total sleep duration and, 8. sleep quality. In parameters 1 to 7, the respondent responds in terms of duration (hours or minutes). In question 8, he/she gives a score between 1 and 6. 1: very poor 6: very good. The higher the score, the better the sleep quality. It was used to measure the change in sleep-related problems of infants in the intervention group at 8 weeks. Information was obtained by filling in the information from the parents of the infants.
Investigation of the change in childrens social-emotional development with Vineland Social-Emotional Early Childhood Scale (VSEES) in the intervention group receiving Snoezelen-Based Occupational Therapy training in 8 weeks | Baseline and Week 8
  Vineland Social-Emotional Early Childhood Scale (VSEES):
  The VSEES is used to assess the social-emotional development of children from birth to 5 years and 11 months. The scale evaluates the interaction/communication dimension, social communication, interest in play, coping and adaptation parameters of infants with its sub-parameters. Score Key: 2=Usually 1=Sometimes 0=Never O= Unlikely B= I don't know. The higher the score, the better the result. It was used to measure the change in social-behavioral problems of infants in the intervention group at week 8. The information was obtained by filling in information from the infants' parents.

CONTACTS AND LOCATIONS:
Locations (1):
- kızılcahamam Health Services Vocational School, Ankara, Kızılcahamam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want the results to be interpreted

REFERENCES:
- [Background] Anderson K, Bird M, Macpherson S, McDonough V, Davis T. Findings from a pilot investigation of the effectiveness of a snoezelen room in residential care: should we be engaging with our residents more? Geriatr Nurs. 2011 May-Jun;32(3):166-77. doi: 10.1016/j.gerinurse.2010.12.011. Epub 2011 Feb 9. PMID 21306798
- [Background] Bishir M, Bhat A, Essa MM, Ekpo O, Ihunwo AO, Veeraraghavan VP, Mohan SK, Mahalakshmi AM, Ray B, Tuladhar S, Chang S, Chidambaram SB, Sakharkar MK, Guillemin GJ, Qoronfleh MW, Ojcius DM. Sleep Deprivation and Neurological Disorders. Biomed Res Int. 2020 Nov 23;2020:5764017. doi: 10.1155/2020/5764017. eCollection 2020. PMID 33381558
- [Background] Krakowiak P, Goodlin-Jones B, Hertz-Picciotto I, Croen LA, Hansen RL. Sleep problems in children with autism spectrum disorders, developmental delays, and typical development: a population-based study. J Sleep Res. 2008 Jun;17(2):197-206. doi: 10.1111/j.1365-2869.2008.00650.x. PMID 18482108
- [Background] Mazurek MO, Sohl K. Sleep and Behavioral Problems in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Jun;46(6):1906-1915. doi: 10.1007/s10803-016-2723-7. PMID 26823076
- [Background] Reynolds AM, Malow BA. Sleep and autism spectrum disorders. Pediatr Clin North Am. 2011 Jun;58(3):685-98. doi: 10.1016/j.pcl.2011.03.009. PMID 21600349
- [Background] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866